CLINICAL TRIAL: NCT05469711
Title: A Study to Determine the Impact Gamification of Routine Airway Clearance Has on the Quality of Life for Children and Young People With Cystic Fibrosis
Brief Title: PlayPhysio: Making Physio Fun
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 295971
Record Dates: First submitted 2021-10-08; First posted 2022-07-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis in Children

STUDY DESIGN:
Intervention Model Description: The study is a single centre, randomised control study with open label participation. Subjects will be randomised 1:1 to either Arm 1 - active arm or Arm 2 - control arm. The trial will last for 4 months 112 days). The first month will be used as a run in period to gather adherence data on both groups with no games available on any of the devices. The gamification will be switched on at day 28 for the participants in arm 1. The trial will run for a further 84 days with the mid-point review half way through this section of the trial.
  Arm 1: intervention-Pp plus gamification Arm 2: control- Pp only - Pp acting as adherence monitor only with no feedback given in real time to patient.
Who Masked: Investigator
Masking Description: Subjects will receive notification to their device on day 1 of the run in period informing them of their group allocation Investigators (PI and CI) will be blinded as to patient allocation. Sub-investigator will be familiar with Playphysio device and will NOT be blinded. This investigator will not be involved in recording of any data but will be available to assist with technical issues faced by patients and provide standard clinical reviews.
  Statistician will be blinded to group allocation Playphysio team will not be blinded and will be able to assist with Playphysio queries that arise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: (Experimental): Gamification
  Interventions: Device: PlayPhysio
- Arm 2 (No Intervention): Monitoring

INTERVENTIONS:
Device: PlayPhysio — The gamification will be switched on at day 28 for the participants in arm 1. The trial will run for a further 84 days with the mid-point review half way through this section of the trial.
  Arms: Arm 1:

SUMMARY:
A study to examine if the gamification of routine airway clearance can improve the quality of live for young people living with chronic health conditions.

DETAILED DESCRIPTION:
CF experts agree that there is a discrepancy between objective and self-reported adherence. Thus, an intervention focusing on both long-term, sustainable monitoring as well on enhancing and sustaining an efficient rate of respiratory physio is urgently needed. The device under investigation here is devoted exactly to this twofold task. Playphysio®(Pp) is a gamification system developed by Will Jackson, who has a background in product and software design but more importantly is the father of an adolescent girl with CF. The Pp is an electronic monitor which can be attached to the outside of an OPEP device. It senses patients' use of the OPEP device to enable the individual completing their existing airway clearance therapy to play mobile games throughout their treatment. Pp enables the individual to pick from a number of games to play whilst completing their normal prescribed airway clearance treatment. The games have been designed so that the ideal treatment technique is encouraged and the individual's treatment routine is supported with the counting of treatment breaths and prompting a pause to carry out their FET and cough. The aim of Pp is to enhance treatment adherence through its innovative element: gamification. It also offers objective monitoring of CF physio adherence through its technology. The Pp app offers positive feedback following the completion of treatment sessions, keeps a record of treatments done and shares this information with the CF physiotherapy team.

A previous study of an earlier Pp device have found good adherence over a 24 week period, however only 17/30 participants completed the trial. Qualitative data found positive outcomes with 2 participants making the following observations. This was an earlier prototype and changes have been made since that time to both the device and the games.

"I rely on the Playphysio for breathing into his PEP device properly. I can't imagine having to go back to the continuous monitoring and timing that used to be required before having Playphysio®" "I rely on Playphysio®. it has reduced my stress and time to get him to do it properly".

Children with CF who are using a play physio device, compared with those not using a play physio, will have a better experience of airway clearance leading to improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

Subject has confirmed diagnosis of cystic fibrosis as determined by the investigator Under care of Alder Hey Cystic Fibrosis Team (local or network care) Subjects 6 years-11 years, 8 months of age, inclusive, on the date of the informed consent Using a compatible OPEP device for daily airway clearance

Exclusion Criteria:

Incompatible device for airway clearance Outside of recruiting age

Ages: 72 Months to 140 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-11 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | Duration of study (4 months)
  This external pilot open randomised controlled trial will generate data examining study feasibility and specifically data on accrual, adherence and outcome measure stability. It is anticipated that data collected will inform power calculations for a future randomised controlled trial. The aim of this subsequent definitive study will be to determine whether Playphysio® with gamification in children with CF is more effective than standard therapy in improving adherence and quality of life. The pilot trial will also be used to gain experience about the use and the satisfaction of the Pp device among young patients.

SECONDARY OUTCOMES:
Cystic Fibrosis Questionnaire-Revised (CFQ-R) | Duration of study (4 months)
  This is a disease-specific health-related quality of life (HRQOL) measure and the relevant measure. An change in score indicating improved quality of life would be a positive outcome. Score range = 0-100 and a higher score indicates higher health related quality of life.
Patient Satisfaction | Duration of study (4 months)
  Questionnaire - an demonstration of high patient satisfaction would be a positive outcome.
Spriometry | Duration of study (4 months)
  Lung function as performed for clinical practice (FEV1 and FVC)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Walsh, BSc, Principal Investigator — Clinical Specialist Physiotherapist in Cystic Fibrosis
Locations (1):
- Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No